CLINICAL TRIAL: NCT00591929
Title: Use of Continuous Passive Motion in the Post-Operative Treatment of Intra-articular Knee Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Collaborators: Orthopaedic Trauma Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GHS-12-06-03
Record Dates: First submitted 2007-12-28; First posted 2008-01-11 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Intra-articular Knee Fractures
MeSH Terms: interventions — Motion Therapy, Continuous Passive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): No Continuous passive motion following ORIF of fractures around the knee
- 2 (Active Comparator): Continuous Passive Motion following ORIF of fractures around the knee
  Interventions: Other: Continuous Passive Motion

INTERVENTIONS:
Other: Continuous Passive Motion — at least 48 hours of continuous passive motion following ORIF of fractures around the knee
  Arms: 2

SUMMARY:
Decreased range of motion is common after fractures around the knee and can impact a patient's ability to perform activities of daily living such as rising from a seated position or getting in and out of a bathtub. A continuous passive motion (CPM) machine is a machine that continuously moves a joint (such as the knee) without the patient having to use the muscles in his/her leg. A goal of this therapy is to maintain as much motion as possible following this injury. This study is a randomized, prospective study to evaluate the effectiveness of CPM in maintaining knee range of motion following open reduction and internal fixation (ORIF) of fractures around the knee

ELIGIBILITY:
Inclusion Criteria:

* If the patient has an intra-articular distal femur or proximal tibia fracture
* Independent ambulatory prior to injury
* No previous knee injury limiting motion

Exclusion Criteria:

* If the patients range of motion was decreased prior to injury (ex. Osteoarthritis, previous knee fracture or injury)
* Any contraindication to CPM (concomitant hip or ankle fracture)
* Open physis of tibia or distal femur
* Pathological Fracture
* Compartment Syndrome
* Neurovascular injury
* Fracture due to gunshot wound
* Greater than 21 days from fracture to definitive open reduction and internal fixation
* Fractures treated with definitive external fixation
* Open fractures
* Extensor mechanism injuries
* Likely problems in the judgment of the investigator with maintaining follow-up

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-12; Primary Completion 2012-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Knee Range of Motion | 48 hours, 2 weeks, 6 weeks, 3 months, 6 months and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kyle J. Jeray, MD, Principal Investigator — Greenville Hospital System
Locations (1):
- Greenville Hospital System Univeristy Medical Center, Greenville, South Carolina, United States